CLINICAL TRIAL: NCT01245582
Title: A Randomized Phase III Study of Oxaliplatin (Eloxatin) and Capecitabine on Top of Sorafenib Versus Sorafenib Alone as First-line Palliative Treatment in Advanced Hepatocellular Carcinoma Patients
Brief Title: Oxaliplatin and Capecitabine on Top of Sorafenib Versus Sorafenib Alone in Advanced Hepatocellular Carcinoma Patients
Acronym: SECOX
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11719; U1111-1115-8557 (Other: UTN); OXALI_R_05123 (Other: sanofi-aventis other reference)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Hepatic Neoplasm Malignant
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Capecitabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SECOX regimen (Experimental): Oxaliplatin (Eloxatin) 85mg/m2 , 2 hour infusion, day 1 Capecitabine (Xeloda) 850 mg/m2 BID orally daily, from day 1 to 7 Sorafenib (Nexavar) 400 mg BID orally daily, from day 1 to 14 (continuously)
  Interventions: Drug: oxaliplatin (SR96669); Drug: capecitabine; Drug: sorafenib
- Sorafenib alone (Active Comparator): Sorafenib (Nexavar) 400 mg BID orally daily, from day 1 to 14 (continuously)
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: oxaliplatin (SR96669) — Pharmaceutical form:injection
  Route of administration: intravenous
  Arms: SECOX regimen
Drug: capecitabine — Pharmaceutical form:tablet
  Route of administration: oral
  Arms: SECOX regimen
Drug: sorafenib — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the efficacy of SECOX regimen by adding oxaliplatin plus capecitabine to sorafenib versus sorafenib alone as palliative treatment for unresectable HCC patients to prolong overall survival (OS) for advanced HCC patients.

Secondary Objective:

* To compare the efficacy of SECOX regimen with Sorafenib alone for progression free survival (PFS)
* To compare the efficacy of SECOX regimen with Sorafenib alone for response rate (RR)
* To assess the overall safety profile of SECOX regimen in comparison of Sorafenib alone

DETAILED DESCRIPTION:
For each patient, the study consists of a baseline period of screening up to 2 weeks, a treatment period with 2 weeks as one study treatment cycle.

Each patient will be randomly assigned to receive either SECOX (Sorafenib, Oxaliplatin with Capecitabine) or Sorafenib alone every 2 weeks until disease progression, intolerable toxicity, or patient's refusal of further study treatment. There will be a 30-day follow-up visit after the last study treatment.

All patients will be follow-up every 2 months until death is observed during post-treatment follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Subjects with histologically or cytologically or clinically diagnosed advanced HCC not amenable to surgical or local treatment. Documentation of original pathology for diagnosis is acceptable if tumor tissue is unavailable at screening.
* Signed written informed consent

Exclusion criteria:

* Clinically diagnosed subjects who did not meet two following criteria:

  * cirrhotic patients with focal lesion > 2cm with arterial hypervascularization demonstrated by 2 coincident imaging techniques
  * cirrhotic patients with focal lesion > 2cm with arterial hypervascularization demonstrated by 1 imaging technique and associated with Alpha Fetoprotein (AFP) level > 400 ng/mL
* Subjects who are receiving or previously received any other investigational therapy or any other systemic anti-cancer treatment for HCC including chemotherapy, immunotherapy or targeted agents, except radiotherapy to non-target lesion (bone metastasis, etc) and HCC adjuvant therapy which was completed more than 6 months prior to randomization. Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior to randomization.
* Subjects with main portal vein thrombosis.
* Subjects with encephalopathy or history of encephalopathy, ascites uncontrolled by medication, active or history of variceal or gastrointestinal bleeding within 30 days
* Subjects with Central Nervous System (CNS) metastasis
* Subjects without one target tumor lesion that be measurable at baseline according to Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria
* Subjects who have received local therapy such as surgery, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection within 4 weeks prior to randomization
* Subjects with Child-Pugh > A
* Eastern Cooperative Oncology Group (ECOG) > 2
* Subjects with inadequate bone marrow, liver and renal function
* Subjects with previous liver transplantation
* Subjects with other serious diseases or medical conditions within 6 months that might be associated with a life expectancy of less than 3 months
* Subjects with other malignant disease previously or concurrently, except cured basal cell carcinoma of skin, cervical carcinoma in situ or any cancer curatively treated > 3 years prior to study entry
* Subjects with known severe hypersensitivity to sorafenib or any other component of sorafenib
* Pregnant or lactating women, or women of child bearing potential without contraceptive method or unwilling to take effective contraception during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of randomization to the date of death due to any cause.
  defined as the time from randomization to the date of death due to any cause. If death is not observed at the cut off date, data on OS will be censored at the last date when patient is known to be alive or the cut-off date, whichever comes first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the date of randomization to the date of documentation of progression or death.
  defined as the time interval from the date of randomization to the date of first observation of disease progression or the date of death (due to any cause). If death or progression is not observed, data on PFS will be censored at the earlier date of last tumor assessment without evidence of progression and the cut-off date.
Response Rate (RR) | From the date of randomization to the end of study.
  defined as the proportion of patients with confirmed complete response (CR) or confirmed partial response (PR), defined by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi